CLINICAL TRIAL: NCT06454760
Title: Risk Factors and Frequency of Acute Idiopathic Hepatitis in Children at Assiut Children Hospital
Status: Not yet recruiting | Type: Observational
Sponsor: Youssef Khalifa Fakher Botros (Other)
Responsible Party: Sponsor-Investigator, Youssef Khalifa Fakher Botros, Resident doctor in pediatric department, Assiut University
Organization: Assiut University (Other)
Other Study IDs: Acute idiopathic hepatitis
Record Dates: First submitted 2024-05-27; First posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Risk Factors and Frequency of Acute Idiopathic Hepatitis in Children at Assiut Children Hospital
Keywords: Hepatitis
MeSH Terms: conditions — Hepatitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. Determine the predisposing factors of acute hepatitis caused by heptotropic and non-hepatotropic viruses in children attending Assiut Children Hospital .
2. Determine the frequency of acute hepatitis caused by hepatotropic and non-hepatotropic viruses in children attending Assiut Children Hospital

DETAILED DESCRIPTION:
* Acute hepatitis has a wide range of repercussions. It can clear up completely and course without any symptoms and without the patient noticing its presence, but in some instances, it can also have complications, in which case it is classed as severe hepatitis. In these cases, the patient suffers from liver failure. The inflammation causes the liver to stop functioning correctly and coagulation disorders arise, which can evolve into hepatic encephalopathy (drowsiness, stupor, disorientation) and even hepatic coma.
* In some cases, infection persists over time and develops into chronic hepatitis, which is when the inflammation of the liver lasts for more than 6 months. Chronic hepatitis can evolve into fibrosis (when the liver cells are inflamed they produce a more fibrous tissue similar to scarring) and eventually cirrhosis (which is when the liver is so damaged and full of scar tissue that it progressively suffers a loss of function) or liver cancer.
* Recent reports of acute hepatitis of unknown origin in previously healthy children have been increasing worldwide. The main characteristics of the affected children were jaundice and gastrointestinal symptoms. By May 2022, the outbreak had affected over 800 children under the age of 16 years in more than 40 countries, resulting in acute liver failure in approximately 10%, including at least 21 deaths and 38 patients requiring liver transplantation.
* Hepatitis is an inflammation of the liver that can be caused by viral infections, alcohol consumption, toxins, medications, and certain other medical conditions. So far, the cause of these cases is unknown, and many hypotheses remain open, but hepatitis AE viruses have been ruled out.

COVID-19 vaccines have also been ruled out, as most of the children are too young and had not been vaccinated. Other possible causes, including other types of coronaviruses, other infections, or environmental causes, are being actively investigated. At this stage the role of the viruses found in some of the cases in the hepatitis pathogenesis is still unclear. No other clear epidemiological risk factors have been identified to date, including recent international travel.

* There was still no confirmed cause, although there were several different working hypotheses, such as severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), adenovirus serotype 41, or SARS-CoV-2 superantigen-mediated immune cell activation. Here, review early observations of the 2022 outbreak which may inform diagnosis.

The clinical syndrome in all identified cases was acute hepatitis with markedly elevated liver enzymes. Many cases reported gastrointestinal symptoms including abdominal pain, diarrhea, and vomiting that preceded presentation with severe acute hepatitis, elevated liver enzyme levels (aspartate transaminase (AST) or alanine aminotransaminase (ALT) > 500 IU/L) and jaundice. Most cases did not have fever.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 1year to 16 years who presented with acute hepatitis were included in the study

Exclusion Criteria:

* Patients with liver cirrhosis
* patients withliver fibrosis
* patients with hepatic cell failure
* patients with hepatic malignancy.

Ages: 1 Year to 16 Years | Sex: All
Age Groups: Child
Study Population: All children aged 1year to 16 years who presented with acute hepatitis were included in the study, and then they will be classified according to the etiology, to detect the frequency of cases with acute idiopathic hepatitis.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Body mass index observation | for about two weeks after recovery from the acute attack
  We will observe the body mass index based on the weight and height of the child and compare that with the previous results before the attack ...for a period of two weeks after recovery.
  2_Determine the frequency of acute hepatitis caused by hepatotropic and non-hepatotropic viruses in children attending Assiut Children Hospital

REFERENCES:
- See also: Related Info — https://www.who.int/emergencies/disease-outbreak-news/item/2022-DON376
- See also: Related Info — https://www.who.int/emergencies/disease-outbreak-news/item/DON-389